CLINICAL TRIAL: NCT04833712
Title: Stereotactic Radioablation for the Treatment of Refractory Atrial Fibrillation
Acronym: RAD-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Spyridon Deftereos, Professor, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 517/17.9.2020
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Arrythmia; Cardiovascular Diseases; Heart Arrhythmia
Keywords: AF
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Radioablation (Experimental): Noninvasive Stereotactic Radioablation will be delivered in a single fraction to electrical isolate the pulmonary veins under CT-guidance.
  Pulmonary vein isolation will be assessed by using Cardioinsight non-invasive mapping system
  Interventions: Radiation: Stereotactic Radioablation

INTERVENTIONS:
Radiation: Stereotactic Radioablation — Stereotactic Radioablation targets on the pulmonary vein ostium aiming to achieve PVI

SUMMARY:
The study aims to investigate the short-term (3 months) and intermediate-term (12 months) safety and preliminary efficacy of stereotactic radiotherapy for pulmonary vein isolation to treat refractory atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia. Current guidelines recommend catheter ablation of AF in symptomatic patients refractory to antiarrhythmic therapy. Pulmonary vein isolation (PVI) remains the cornerstone of any ablation procedure irrespective of patient characteristics. Recently, single fraction stereotactic radioablation has been used in patients with ventricular arrhythmias non-eligible for transcatheter ablation or after a failed transcatheter ablation.

This is a single center, single arm, prospective and phase 1 clinical trial. Patients with refractory AF non-eligible for transcatheter ablation or after a failed transcatheter ablation will receive stereotactic radioablation for PVI.

The target contours for paroxysmal AF stereotactic radioablation will cover the left atrial-venous wall, the myocardium and the myocardial sleeves of the PVs transmural at the PV antrum, similar to catheter ablation. The contours will be approximately 4-6 mm wide along the PVs / LA and approximately 2-4 mm deep depending on the tissue thickness.

A pre-validation study will evaluate the location with respect to right and left PVs. Patients with esophagus in direct contact with the actual target lesion will be excluded.

PVI will be assessed by means of Cardio Insight non invasive mapping system during radioablation.

Safety is the primary endpoint of the study. Safety will be assessed by incidence and evaluation of any serious adverse evens using CTCAE V5.0 criteria associated with the procedure through 90 days (short-term) and 12 months (intermediate term).

Efficacy will be evaluated by assessing atrial fibrillation recurrence and AF burden after 90 days of blank period until 12 months post-treatment based on pacemaker interrogation.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-89
* Paroxysmal or persistent symptomatic AF refractory to antiarrhythmic drugs.
* Failure from the previous catheter ablation of AF, or contraindicate /unwilling to undergo catheter ablation.
* Dual chamber pacemaker implanted
* Understands the nature of the study, treatment procedure and provides written informed consent
* Willing to comply with specified pre-, post- and follow-up testing, evaluations and requirements

Exclusion Criteria:

* Permanent AF
* Unstable angina
* Presence of any disease that is likely to shorten life expectancy to < 1 year
* Any cardiac surgery within three months prior to enrolment
* Awaiting cardiac transplantation or other cardiac surgery within the next year
* Myocardial infarction (MI) within 60 days prior to enrolment
* Contraindications to oral anticoagulation
* Active systemic infection or sepsis
* History of a documented thromboembolic event such as stroke or transient ischemic neurological attack (TIA) in the three months prior to enrollment.
* Any other clinical condition that might jeopardize patient safety during participation in this trial or prevent the subject from adhering to the trialprotocol
* Esophageal ulcer.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-10 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
90 days adverse events by CTCA5 | 90 days
  Safety will be assessed by incidence and evaluation of any adverse events using CTCA5 V5.0 criteria that are related to the procedure

SECONDARY OUTCOMES:
12 months adverse events by CTCA5 | 12 months
  Safety will be assessed by incidence and evaluation of any adverse events using CTCA5 V5.0 criteria that are related to the procedure
Recurrence of atrial fibrillation after 90 days blanking period post-treatment | 90 days
Atrial fibrillation burden reduction after 90 days blanking period post-treatment | 90 days to 12 months
Cardiovascular Mortality | 12 months
All-Cause Mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Attikon University Hospital, Chaïdári
  - Mediterraneo Hospital, Glyfada

IPD SHARING:
Plan to Share IPD: No